CLINICAL TRIAL: NCT05612620
Title: Elucidating the Microbiome in Patients With Recurrent Pregnancy Loss Vs. Patients Without Gynecological or Obstetrical Conditions
Brief Title: Elucidating the Microbiome in Patients With Recurrent Pregnancy Loss
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assuta Ashdod Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 0140-21-AAA
Record Dates: First submitted 2022-10-23; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-09

CONDITIONS: Microbiome; Recurrent Pregnancy Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Samples from uterine discharge vaginal discharge and stool samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RPL: Samples from the vagina, fornix and cervical canal and rectum will be taken by introducing a flocked nylon swab to the vagina via a speculum and circular swabbing for 5-10 seconds before using any antiseptics.
  Interventions: Diagnostic Test: coulture
- Healthy: Samples from the vagina, fornix and cervical canal and rectum will be taken by introducing a flocked nylon swab to the vagina via a speculum and circular swabbing for 5-10 seconds before using any antiseptics.
  Interventions: Diagnostic Test: coulture

INTERVENTIONS:
Diagnostic Test: coulture — Samples from the vagina, fornix and cervical canal will be taken by introducing a flocked nylon swab to the vagina via a speculum and circular swabbing for 5-10 seconds before using any antiseptics.

SUMMARY:
Recurrent pregnancy loss (RPL) is defined as 2 or more consecutive miscarriages1 This condition affects about 1-3% of couples during their reproductive years. The role of vaginal infections in RPL is controversial and microbiological screening is not recommended as per the international guidelines. Current theories suggest that altered vaginal and uterine microbiota may trigger an inflammatory response in the endometrium even without the presence of clinical infection which could affect the success of embryo implantation and future development of pregnancy2 .Changes in the uterine microbiota can lead to chronic endometritis (CE). This condition is caused by continuing inflammation of the endometrium, involving a variety of common bacterial and yeast species and has been associated with RPL3 . Notably, CE can be found in up to 45% of infertile patients4. Current diagnosis of CE is based on histopathological examination, immunohistochemistry assay for CD138 cells and morphological appearance on hysteroscopy. While antibiotic treatment can improve ongoing pregnancy rates in patients with RPL treatment success is still partial and unpredictable. A mechanistic link is yet to be established between vaginal and uterine microbiota and RPL and it is unknown whether restoration of the microbiome in patients with RPL can improve pregnancy outcomes.

DETAILED DESCRIPTION:
Aims The aim of the current study is to evaluate vaginal and intrauterine microbiota in women with recurrent pregnancy loss (RPL) as compared to normal controls. Ultimately we would like to assess whether women with RPL have a characteristic microbiome which may be significantly different microbiota of healthy patients in our study population. This could later lead to treatment with a tailored microbiota transplantation approach involving healthy vaginal microbiota for the treatment of patients with RPL and implement it in a prospective randomized controlled trial in order to modulate the reproductive tract microbiota and achieve and improved pregnancy outcome.

Background

A rapidly growing field in biologic research of human health and disease is that of microbiome research. The microbiome inhabiting the female reproductive tract has long been suspected to play an important role in health and disease. Current theories suggest that altered microbiota even without clinical infection may trigger an inflammatory response in the endometrium. It affects the success of embryo implantation and future development of pregnancy.5 Most studies deal with genital tract microbiome in patients with repeated implantation failure in IVF, however, some studies have also found altered microbiome in patients with recurrent pregnancy loss (RPL)6 Vaginal and endometrial microbiotas might be independent. Endometrial microbiota has a richer alpha diversity than vaginal microbiota, and dysbiosis of vaginal or endometrial microbiota can cause implantation failure. Unlike previous reports, Ichiyama et al reports that the Lactobacillus rate in the vagina, but not the endometrium, may be a biomarker for repeated implantation failure7 Small studies showed association between spontaneous abortion and abnormal vaginal microbiome( 60% intermediate flora, 20% BV condition), with higher levels of selected metabolites in the vaginal environment (e.g., inosine, fumarate, xanthine, benzoate, ascorbate)8 Recurrent pregnancy loss (RPL) is defined American Society for Reproductive medicine as two or more spontaneous miscarriages before gestational week 22 (not necessarily consecutive) The role of vaginal infections in RPL is controversial and screening for infections is not routinely recommended in patients with RPL9

Major immune cells in the human endometrium include uterine Natural Killer (uNK) cells, macrophages, dendritic cells (DCs) and T cells. Each of these cell populations demonstrated a specific role. uNK are involved in the success of implantation and maintenance of pregnancy through their ability both to interact through inhibitor receptors with HLA-G, HLA-E and HLA-C expressed on trophoblast cells and to produce angiogenic factors Kuon et al in their small study described that RPL patients with elevated pNK suffer more often from colonization by Gardnerella vaginalis and gram-negative anaerobes . This might indicate an association between the vaginal microbiota, local inflammation, changes in immune parameters and miscarriage.10 Like the vaginal microbiome, the endometrial microbiome is usually dominated by Lactobacilli. 11 A recent studies illustrated that the presence of a non-Lactobacillus-dominating microbiome in endometrial fluid of IVF patients was associated with significantly lower implantation, pregnancy and live birth rates 12 13 According to researches microbiota composition in endometrial fluid does not fully reflect that in endometrial tissue.14 However, only few studies have directly probed the microbes within the uterine environment and how these microbes could influence in implantation , the majority of them in IVF cycles.

First trimester miscarriage can be associated with reduced prevalence of Lactobacillus spp. and with changes in the relative abundance of several bacterial genera, including Fam_Finegoldia, Lac_Coprococcus_3, and Lac_Roseburia 15 16

Chen W et al showed the relative abundances of Actinobacteria and Fusobacteria in the so called Chronic endometritis group at the phylum level.At the genus level, high relative abundances of Gardnerella were observed in the Chronic endometriosis and non-pregnancy groups, which significantly referred to the negative IVF outcome17

Settings and participants All patients referred to Assuta Ashdod university hospital due to RPL, meeting the inclusion criteria, will be offered recruitment.

Inclusion criteria include:

• women aged 18-40 years old, with two or more consecutive miscarriages.

Exclusion criteria will include:

* documented past PID,
* previous history of uterine malformations,
* patients with hyperplasia and endometrial cancer,
* patients with IUD and antimicrobial treatment in the preceding 4 weeks.

Study methodology and techniques

Study design

After obtaining informed consent we will collect samples from 4 anatomical locations: lower third of vagina (before speculum placement), posterior fornix and cervical canal ( after sterile speculum placement), and a sample of gut microbiome.

Sample size - 20 women for each pathology in the research group and 20 women control group, this is similar to other studies on the subject 4.

The following data will be collected from medical records:

* age,
* ethnicity,
* BMI,
* Lifestyle: tobacco use, Number of partners in the past 6 months, diet, hygienic procedures,
* Gynecological and obstetrical history: gravidity, parity, menarche time, regularity of menstrual cycle,
* Type and duration of contraception,
* Symptoms: pain, menometrorrhagia,
* Sonographic findings,

Samples from the vagina, fornix and cervical canal will be taken by introducing a flocked nylon swab to the vagina via a speculum and circular swabbing for 5-10 seconds before using any antiseptics. Thus a total of 160 samples (3 patients groups (n=20*2) * 4 samples) will be taken.

Samples will be snap frozen at -80c and kept until further analysis. Batched swab specimens will undergo microbial DNA extraction using standard protocols of the Human Microbiome Project (HMP). Following extraction, a PCR reaction for 16S RNA gene amplification will be performed using HMP primers sets. 16S amplicons will be sequenced using an Illumina next-generation sequencing platforms (PE 250bpX2).

Sequencing data will be analyzed at the Moran-Gilad lab, Ben-Gurion University. The bioinformatics analysis will be based on the QIIME software package pipeline18 . Briefly, microbiome data will be analyzed using standard methods for rarefaction, alpha and beta diversity and abundance of taxa at different taxonomical levels. The ANOVA test will be used to determine if OTU relative abundance is different between samples, the G test of independence will be used to determine association of OTU presence/absence with a specific category, and significant variation between sample groups will be analyzed using DESeq2 R package 19on the raw non-normalized OTU biom table.

Recruitment strategy

Patients will be recruited from outpatients clinic at the Samson Assuta University Hospital in accordance with a protocol that is under approval process of the local Institutional Review Board (IRB).

The investigator will inform the patient about the study, its purpose, and method of randomization of study groups. Patients will not be cajoled into participating in this study. The Investigator will discuss foreseeable risks involved, as well as potential benefits, for each study group. Patients who have consented to having their information obtained during the study for analysis of the results will have their confidentiality maintained at all times using a study code as an identifier in the research database. The patients will be informed by the Investigator that their medical treatment will not be affected in any mean by their decision whether to participate or not in the study. Patients will be informed that they may choose to withdraw from the study at any stage without jeopardizing any further medical care. A signed and dated Informed Consent must be obtained by the Investigator from the patient prior to enrolment into this study. The original signed and dated information sheet and patient consent will be kept by the Investigator. A signed copy will be provided to the patient.

Statistical analysis

Statistical analysis will be performed using R software environment for statistical computing and graphics. Categorical variable data will be presented using percentile and statistical significance will be tested using the X² or Fisher's exact test, as appropriate. Ordinal variable data will be presented using median and inter quartile range and statistical significance will be analyzed using Mann Whitney test. Continuous variable data will be presented using mean and standard deviation, Student t test will be used for statistical analysis

Ethics

This study protocol will be submitted to Assuta Ashdod University Hospital Ethics committee for approval. The study will be conducted in accordance with the ethical principles originating from the Declaration of Helsinki and GCP (ICH E6) and in compliance with local regulatory requirements. Participants' identity will be kept confidential, and to the extent permitted by the applicable laws and/or regulations, will not be made publicly available. If the study results are published, the participants' identity will remain confidential.

Informed consent will be obtained in accordance with ICH/GCP Guidelines and the Declaration of Helsinki and will be implemented before protocol specific procedures are carried out. The risks and benefits of participating in the study will be verbally explained to each potential participant prior to signing the consent form in accordance with local regulatory legal requirements. The signed consent form will be retained by the investigator and a copy provided to each participant.

Source Documentation

The investigator will keep accurate separate records of all participants' study data collected, including all pertinent study related information. The investigators are committed to thorough documentation of all side effects and Adverse Events during the study in a participant study binder including any diagnostic tests conducted during the study.

All study documentation will be kept for 15 years after all participants have completed and all data has been collected. The IRB/IEC will be notified in writing of the study completion and archive site.

ELIGIBILITY:
Inclusion Criteria:

* • women aged 18-40 years old, with two or more consecutive miscarriages.

Exclusion Criteria:

* • documented past PID,

  * previous history of uterine malformations,
  * patients with hyperplasia and endometrial cancer,
  * patients with IUD and antimicrobial treatment in the preceding 4 weeks.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with two or more consecutive miscarriages ages 18-40 With a normal uterine cavity as per hysteroscopy, no chromosomal abnormalities and negative APLA test.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-11-14 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Microbiome differences in patients with repeat pregnancy loss and healthy population | through study completion, an average of 2 years
  microbiome data will be analyzed using standard methods for rarefaction, alpha and beta diversity and abundance of taxa at different taxonomical levels. A statistical analysis will be performed in order to evaluate if there is a significant difference in the presence of different bacteria strains in patients with a history of RPL and healthy controls

CONTACTS AND LOCATIONS:
Overall Officials: Oshri Barel, MD, Principal Investigator — Assuta Ashdod Hospital
Locations (1):
- Assuta Ashdod University Hospital, Ashdod, Israel